CLINICAL TRIAL: NCT05217238
Title: Median Effective Dose of Remifentanil for the Prevention of Pain Caused by the Injection of Rocuronium
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Zhuan Zhang, Director, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20211218
Record Dates: First submitted 2021-12-18; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Rocuronium; Injection Pain
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Age range of 18 to 44 years olds (Experimental): The initial dose of lidocaine for pre-injection was set at 1ug/kg according to previous literature and preliminary test results. The dose of remifentanil was according to the patients' pain level. If there is no pain (negative reaction), the dose of remifentanil in the next patient will be reduced until the patient has pain. If there is pain (positive reaction), the dose of remifentanil will be increased in the next patient until the patient is painless.
  Interventions: Drug: Remifentanil
- Age range of 45 to 59 years olds (Experimental): The initial dose of lidocaine for pre-injection was set at 1ug/kg according to previous literature and preliminary test results. The dose of remifentanil was according to the patients' pain level. If there is no pain (negative reaction), the dose of remifentanil in the next patient will be reduced until the patient has pain. If there is pain (positive reaction), the dose of remifentanil will be increased in the next patient until the patient is painless.
  Interventions: Drug: Remifentanil
- Age range of 60 to 80 years olds (Experimental): The initial dose of lidocaine for pre-injection was set at 1ug/kg according to previous literature and preliminary test results. The dose of remifentanil was according to the patients' pain level. If there is no pain (negative reaction), the dose of remifentanil in the next patient will be reduced until the patient has pain. If there is pain (positive reaction), the dose of remifentanil will be increased in the next patient until the patient is painless.
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — Advanced intravenous injection of remifentanil before the rocuronium injection

SUMMARY:
As a medium-and long-term non-depolarizing muscle relaxant, rocuronium has the advantages of quick effect, no histamine release and accumulation and no obvious cardiovascular adverse reactions, so it has been widely used in clinical anesthesia induction. However, when given intravenously, rocuronium can cause adverse reactions such as injection pain and limb retraction, which can lead to needle prolapse, extravasation of injection drugs, swelling of injection site, serious induction delay, and cardiovascular adverse events in severe cases. Remifentanil is a synthetic opioid drug hydrolyzed by esterase. Compared with other opioid drugs, remifentanil has the advantages of quick effect, short half-life and short time of hemodynamic changes, so it is an ideal analgesic in clinical anesthesia. In this study, in order to provide clinical references, sequential method was used to find the median effective dose (ED50) by means of pre-intravenous injection of Remifentanil to suppress pain in rocuronium injection.

ELIGIBILITY:
Inclusion Criteria:

1. Ages ranged from 18 to 80.
2. ASA # or # level.

Exclusion Criteria:

* Allergy or contraindication to remifentanil or rocuronium; required for Central venipuncture catheterization;
* Abnormal liver or kidney function;
* Heavy drinking and long-term use of sedatives, analgesics or anti-anxiety drugs;
* Hearing and language impairment;
* Peripheral vascular disease;
* Severe cardiovascular disease or neurological disorders;
* Failure of one-time peripheral venipuncture;
* Infection of hand or wrist skin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-12-18 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
The appearance of intravenous injection pain Yes or No | an average of 2 minutes
  Yes or No

SECONDARY OUTCOMES:
The levels of intravenous injection pain | an average of 2 minutes
  The intravenous injection pain in this study was divided into the following 5 levels according to its severity: level 0: After repeated questioning, the patient did not feel any abnormal sensation; level 1: upon inquiry, the patient felt swelling at the intravenous injection site; Level 2: Upon inquiry, the patient felt pain and had no body movement reaction (facial pain expression, arm withdrawal, tears, etc.); Level 3: Upon inquiry, the patient had pain and body movement reaction.
  Or complain of pain without inquiry; Level 4: the patient has a strong reaction and body movement reaction. Level 2 and above is defined as injection pain.

OTHER OUTCOMES:
If any adverse memory or pain during the induction of general anesthesia | the time one hour after turn into Postanesthesia care unit
  Patients recalled by visual analogue scale (VAS) to assess injection pain level : Mark 0 is painless. Mark 10 is violent pain, The numbers between them was pain of varying degrees.

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Hospital of Yangzhou University, Yangzhou, Jiangsu, China

REFERENCES:
- [Derived] Yan S, Wu H, Yu Y, Li N, Yu L, Wang Y, Li H, Zhang D, Zhang Z. Median Effective Dose of Remifentanil for the Prevention of Pain Caused by the Injection of Rocuronium: An Age-Stratified Study. Pain Ther. 2023 Jun;12(3):683-694. doi: 10.1007/s40122-023-00490-5. Epub 2023 Mar 8. PMID 36884108